CLINICAL TRIAL: NCT02596516
Title: A Comparison of Colonic Bile Acid Content Following Right and Left Colectomies
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Ilan Kent, Medical Doctor, Meir Medical Center
Other Study IDs: MMC-0249-15
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2015-11-06 (Estimated); Status verified 2015-11

CONDITIONS: Colectomy; Bile Acid and Salts

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this study is to evaluate whether there is a difference in the bile acid content in the bowel in patients after right versus left colectomy. There is compelling evidence that patients under going resection of the right colon versus left coolon have a lower polyp detection rate in surveillance colonoscopies. The investigators intend to evaluate feces of patients undergoing left and right colectomies; prior to their surgery and again three and six months aftet the surgery. The investigators plan to compare the content of the different bile acids and to compare the content between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18.
* Patients intended to undergo a colectomy for colonic cancer
* Patients willing and participate and able to sign an informed consent

Exclusion Criteria:

* Age under 18.
* Patients with Inflammatory Bowel Disease (Crohn's, Ulcerative colitis).
* Patients refusing to participate or are unable to understand or sign an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients palnned to undergo colon resection.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-01 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Colonic bile acid content | two years